CLINICAL TRIAL: NCT06016530
Title: Multi-level Molecular Profiling of Stress Exposure Under Standardized Food Intake: A Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Nils Gassen (Other)
Responsible Party: Sponsor-Investigator, Dr. Nils Gassen, Principal Investigator, University Hospital, Bonn
Organization: University Hospital, Bonn (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 084/22
Record Dates: First submitted 2023-08-09; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Stress Related Disorder; Nutrition, Healthy; Metabolism
Keywords: Stress Related Disorders; Nutrition; Metabolism

STUDY DESIGN:
Intervention Model Description: One group; all participants will undergo identical measurements, including: 1) Baseline assessment, 2) Sleep Deprivation, and 3) Dexamethasone Supplementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy participants (Experimental): The study will involve 20 to 30 healthy participants, with approximately 15 females and 15 males. Each participant will undergo three measurements: 1) Baseline assessment, 2) Sleep Deprivation, and 3) Dexamethasone Supplementation.
  The baseline measurement will be the starting point taken before any interventions are applied. It will serve as a control and reference to evaluate the impact of interventions.
  Interventions: Behavioral: Sleep Deprivation; Drug: Dexamethasone Supplementation

INTERVENTIONS:
Behavioral: Sleep Deprivation — During a sleep deprivation period lasting over 36 hours, individual fluctuations of various metabolites will be measured throughout the day (12 hours) for each participant while adhering to a standardized diet. To achieve this, blood samples will be collected and processed into plasma or peripheral blood mononuclear cells (PBMCs).
Drug: Dexamethasone Supplementation — Dexamethasone belongs to the drug class of corticosteroids. It is a synthetic glucocorticoid that activates glucocorticoid receptor (GR) and the hypothalamic-pituitary-adrenal (HPA) axis selectively.
  Following the administration of 1 mg of dexamethasone as a pharmacological stressor, individual fluctuations of various metabolites will be measured throughout the day (12 hours) for each participant under a standardized diet. To facilitate this, blood samples will be collected and processed into plasma or peripheral blood mononuclear cells (PBMCs).

SUMMARY:
Nutrition plays a crucial role in preventing various diseases, including cardiovascular and metabolic conditions. Moreover, it is gaining increasing attention in the context of preventing and treating psychiatric disorders. However, limited knowledge exists concerning the effects of food intake and stress on metabolism over time.

To enhance the understanding of this subject, blood components in healthy volunteers will be examined during a standardized diet, focusing on the interaction between nutrition and stress. Physiological stress will be induced by subjecting participants to sleep deprivation for over 36 hours. Hormonal influences related to the female menstrual cycle are particularly taken into account in female participants.

In conclusion, comprehending these processes can improve the understanding of nutritional physiology and contribute to advancements in clinical practice.

DETAILED DESCRIPTION:
Nutrition is crucial in preventing cardiovascular, metabolic, and other diseases, and its significance in psychiatric disorders is growing. It plays a key role in maintaining health and can be a low-risk, cost-effective therapy in early disease stages.

Observational studies suggest that healthy eating habits, such as the Mediterranean diet, positively affect inflammation markers. However, the exact molecular processes during food intake remain limited to observational studies due to the complexity of involved factors. Moreover, the effects of food intake and stress on metabolism over time are poorly understood.

A comprehensive molecular analysis during a standardized diet is crucial for understanding nutrition's role in disease treatment and advancing nutritional analyses in clinical practice. By utilizing a "multi-omics approach," it becomes possible to study changes in various molecular groups, such as proteins or lipids, and investigate the underlying mechanisms of diseases.

For this purpose, a cohort of 20 to 30 healthy individuals, encompassing around 15 females and 15 males, will be recruited. Initially, all participants will undergo a baseline measurement, profiling their blood components while adhering to a standardized diet. Subsequently, the same participants will be subjected to a physiological stressor involving 36 hours of sleep deprivation. Lastly, the participants will receive dexamethasone as a pharmacological stressor. Throughout these stages, the primary focus centers on examining the interaction between nutrition and stress at a metabolic level.

The main goal of the study is to improve comprehension of the molecular mechanisms associated with food intake and stress, and their impact on metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Present written declaration of consent
* Healthy
* BMI between 18 and 30

Exclusion Criteria:

* Insufficient linguistic communication
* Drug abuse or alcohol dependency
* Smoker
* Hormonal contraception
* Neurological condition or epilepsy in the medical history
* Regular medication except for L-thyroxine or antihistamines
* A known disease of the cardiovascular system, hypertension higher than 160/90mmHg

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Proteomics and Autophagy Processes | Changes will be measured throughout one day between 7 a.m. and 7 p.m. (7 blood withdrawals every two hours; at 7 a.m., 9 a.m., 11 a.m., 1 p.m., 3 p.m., 5 p.m., and 7 p.m.). These measurements will be repeated after the two interventions.
  Change in protein levels of autophagy biomarkers (LC3II & p62) in isolated PBMCs (peripheral blood mononuclear cells) using Western Blotting.

SECONDARY OUTCOMES:
Metabolic Processes | Changes will be measured throughout one day between 7 a.m. and 7 p.m. (7 blood withdrawals every two hours; at 7 a.m., 9 a.m., 11 a.m., 1 p.m., 3 p.m., 5 p.m., and 7 p.m.). These measurements will be repeated after the two interventions.
  Metabolic measurements will be conducted using mass spectrometry, a technique that identifies and quantifies molecules based on their mass-to-charge ratio. The units for these measurements will be expressed in molar concentrations (e.g., µM or mM).
Lipid Profiling | Changes will be measured throughout one day between 7 a.m. and 7 p.m. (7 blood withdrawals every two hours; at 7 a.m., 9 a.m., 11 a.m., 1 p.m., 3 p.m., 5 p.m., and 7 p.m.). These measurements will be repeated after the two interventions.
  Targeted and quantitative analysis by mass spectrometry of changes in plasma lipids. The units for lipid concentrations will be reported in mass units (nmol/mL)
Saliva Cortisol Levels | Changes will be measured throughout one day between 7 a.m. and 7 p.m. (hourly: 7 a.m., 8 a.m., 9 a.m., 10 a.m., 11 a.m., 12 p.m., 1 p.m., 2 p.m., 3 p.m., 4 p.m., 5 p.m., 6 p.m., 7 p.m.) These measurements will be repeated after the two interventions.
  Saliva Cortisol Levels in nmol per Liter (nmol/L) after dexamethasone intake will be evaluated and compared to the control group.
The Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS) | The assessments will be conducted twice: at the beginning before baseline measurements, and again before the final intervention. This approach allows for a comparison between the initial state and the state before the final intervention.
  The Warwick-Edinburgh Mental Well-being Scale (WEMWBS) was developed by researchers to measure the mental well-being of adults. WEMWBS is a 14-item scale covering subjective well-being and psychological functioning. All items are worded positively and address aspects of positive mental health. The scale is scored by summing responses to each item, answered on a 1 to 5 Likert scale. The minimum score is 14 and the maximum is 70.
Pittsburgh Sleep Quality Index (PSQI) | The assessments will be conducted twice: at the beginning before baseline measurements, and again before the final intervention. This approach allows for a comparison between the initial state and the state before the final intervention.
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire assessing sleep quality over a 1-month interval. The measure consists of 19 items, creating 7 components that produce one global score. It takes 5-10 minutes to complete. The global PSQI score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, with lower scores indicating better sleep quality.
Resilience Scale (Wagnild &Young) | The assessments will be conducted twice: at the beginning before baseline measurements, and again before the final intervention. This approach allows for a comparison between the initial state and the state before the final intervention.
  The Resilience Scale is a self-reported 25-item scale to assess overall resilience. A higher score means a better resilience. Scores range from 25 to 175 points.
STROOP test | The changes will be measured every two hours throughout the day between 7 a.m. and 7 p.m. The test will be conducted at 7 a.m., 9 a.m., 11 a.m., 1 p.m., 3 p.m., 5 p.m., and 7 p.m. This testing schedule will be repeated for all the interventions.
  The Stroop test is a cognitive task where participants must name the ink color of words while ignoring the actual word meaning. It measures response inhibition and cognitive flexibility. The measure is typically the time taken to complete the task (in seconds), with higher values indicating worse cognitive performance.
N-Back test | The changes will be measured every two hours throughout the day between 7 a.m. and 7 p.m. The test will be conducted at 7 a.m., 9 a.m., 11 a.m., 1 p.m., 3 p.m., 5 p.m., and 7 p.m. This testing schedule will be repeated for all the interventions.
  The N-Back test is a cognitive task that assesses working memory and attention. Participants are required to indicate whether a current stimulus matches the one presented 'N' steps back in a sequence. Scores are reported as a percentage of correct responses, with higher percentages indicating better cognitive performance.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Department of Psychiatry and Psychotherapy, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
All data will be anonymized, so that no participant will suffer any disadvantage.

REFERENCES:
- [Background] Bastard JP, Jardel C, Bruckert E, Blondy P, Capeau J, Laville M, Vidal H, Hainque B. Elevated levels of interleukin 6 are reduced in serum and subcutaneous adipose tissue of obese women after weight loss. J Clin Endocrinol Metab. 2000 Sep;85(9):3338-42. doi: 10.1210/jcem.85.9.6839. PMID 10999830
- [Background] Berthelot E, Etchecopar-Etchart D, Thellier D, Lancon C, Boyer L, Fond G. Fasting Interventions for Stress, Anxiety and Depressive Symptoms: A Systematic Review and Meta-Analysis. Nutrients. 2021 Nov 5;13(11):3947. doi: 10.3390/nu13113947. PMID 34836202
- [Background] Bowen KJ, Sullivan VK, Kris-Etherton PM, Petersen KS. Nutrition and Cardiovascular Disease-an Update. Curr Atheroscler Rep. 2018 Jan 30;20(2):8. doi: 10.1007/s11883-018-0704-3. PMID 29383458
- [Background] Draper CF, Duisters K, Weger B, Chakrabarti A, Harms AC, Brennan L, Hankemeier T, Goulet L, Konz T, Martin FP, Moco S, van der Greef J. Menstrual cycle rhythmicity: metabolic patterns in healthy women. Sci Rep. 2018 Oct 1;8(1):14568. doi: 10.1038/s41598-018-32647-0. PMID 30275458
- [Background] Estruch R. Anti-inflammatory effects of the Mediterranean diet: the experience of the PREDIMED study. Proc Nutr Soc. 2010 Aug;69(3):333-40. doi: 10.1017/S0029665110001539. Epub 2010 Jun 2. PMID 20515519
- [Background] Hamdy O, Barakatun-Nisak MY. Nutrition in Diabetes. Endocrinol Metab Clin North Am. 2016 Dec;45(4):799-817. doi: 10.1016/j.ecl.2016.06.010. PMID 27823606
- [Background] Leonard BE. Inflammation and depression: a causal or coincidental link to the pathophysiology? Acta Neuropsychiatr. 2018 Feb;30(1):1-16. doi: 10.1017/neu.2016.69. Epub 2017 Jan 23. PMID 28112061
- [Background] Locke A, Schneiderhan J, Zick SM. Diets for Health: Goals and Guidelines. Am Fam Physician. 2018 Jun 1;97(11):721-728. PMID 30215930
- [Background] Marx W, Moseley G, Berk M, Jacka F. Nutritional psychiatry: the present state of the evidence. Proc Nutr Soc. 2017 Nov;76(4):427-436. doi: 10.1017/S0029665117002026. Epub 2017 Sep 25. PMID 28942748
- [Background] Ravera A, Carubelli V, Sciatti E, Bonadei I, Gorga E, Cani D, Vizzardi E, Metra M, Lombardi C. Nutrition and Cardiovascular Disease: Finding the Perfect Recipe for Cardiovascular Health. Nutrients. 2016 Jun 14;8(6):363. doi: 10.3390/nu8060363. PMID 27314382
- [Background] Ridker PM, Buring JE, Cook NR, Rifai N. C-reactive protein, the metabolic syndrome, and risk of incident cardiovascular events: an 8-year follow-up of 14 719 initially healthy American women. Circulation. 2003 Jan 28;107(3):391-7. doi: 10.1161/01.cir.0000055014.62083.05. PMID 12551861
- [Background] Sanner T. Formation of transient complexes in the glutamate dehydrogenase catalyzed reaction. Biochemistry. 1975 Nov 18;14(23):5094-8. doi: 10.1021/bi00694a011. PMID 39
- [Background] Wallace M, Hashim YZ, Wingfield M, Culliton M, McAuliffe F, Gibney MJ, Brennan L. Effects of menstrual cycle phase on metabolomic profiles in premenopausal women. Hum Reprod. 2010 Apr;25(4):949-56. doi: 10.1093/humrep/deq011. Epub 2010 Feb 10. PMID 20150174
- [Background] Watzl B, Kulling SE, Moseneder J, Barth SW, Bub A. A 4-wk intervention with high intake of carotenoid-rich vegetables and fruit reduces plasma C-reactive protein in healthy, nonsmoking men. Am J Clin Nutr. 2005 Nov;82(5):1052-8. doi: 10.1093/ajcn/82.5.1052. PMID 16280438